CLINICAL TRIAL: NCT04238364
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study Followed by a Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability and Pharmacokinetics of EI1071 in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Amount of EI-1071 in Blood in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elixiron Immunotherapeutics (Hong Kong) Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EI1071-001
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: CSF1R Inhibitor; Safety; Tolerability; Pharmacokinetics; EI1071

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EI-1071 Tablet (Experimental): EI-1071 tablet(s) administered orally as single ascending dose(SAD), multiple ascending daily dose(MAD)
  Interventions: Drug: EI-1071
- Placebo (Placebo Comparator): EI-1071 tablet(s) administered orally as single ascending dose(SAD), multiple ascending daily dose(MAD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EI-1071 — EI-1071 Tablet(s)
  Arms: EI-1071 Tablet
Drug: Placebo — Matching Placebo Tablet(s)
  Arms: Placebo

SUMMARY:
This was a first-in-human study to determine the safety, tolerability, and pharmacokinetics of EI1071 after single and multiple doses in healthy volunteers.

DETAILED DESCRIPTION:
This phase 1 first-in-human study was designed to assess the safety, tolerability, and pharmacokinetics of single and multiple doses of EI1071 when administered to healthy adult volunteers. This was a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort trial. The study was conducted in two phases: a single ascending dose (SAD) phase, followed by a multiple ascending dose (MAD) phase. Approximately 58 healthy volunteers enrolled in SAD and MAD cohorts (34 in SAD; 24 in MAD). In SAD, participants in Cohorts 1 to 5 received one dose of EI-1071 or placebo. In MAD, participants in Cohorts 1 and 2 received multiple doses of EI-1071 or placebo for 14 consecutive days. Safety, tolerability, and PK profile of EI-1071 were assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for enrollment in the study only if they met all the following criteria:

1. Healthy male and female subjects, 18 to 45 years of age, inclusive. (Taiwan only: To be at least 20 years of age.)
2. The subject had a body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, and weighs at least 50kg.
3. The subject was in good health and has no medical condition of clinical significance or that may impact the outcome of the study, as determined by the investigator (as determined by medical history, physical examination, 12-lead electrocardiogram [ECG], vital signs, and clinical laboratory results at screening).
4. The subject was able to understand the nature of the study and any potential hazards associated with participating in it.
5. The subject was able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
6. The subject was willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided, and has had the opportunity to discuss the study with the investigator or designee.
7. Negative pregnancy test for female subjects. Women of child bearing potential and Women not of child bearing potential were eligible to participate. Both women of child bearing potential and women of no child bearing potential used an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 90 days after taking the last dose of EI1071). Acceptable methods of contraception included abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method, female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner was surgically sterile or 2 years post-menopausal. All male subjects/partners must agree to consistently and correctly use a condom. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.
8. Subject was currently not using strong inhibitors or inducers of CYP3A4 and was not anticipated to use these for the duration of the study

Exclusion Criteria:

Subjects were eligible for enrollment in the study only if they meet none of the following criteria:

1. The subject had a history of severe allergic or anaphylactic reactions.
2. The subject had a known allergy or hypersensitivity to any component of the formulation.
3. The subject had a medical history or current evidence of any clinically significant (as determined by the investigator) cardiac, endocrine (including diabetes), hematologic, hepatobiliary (abnormal alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transpeptidase [GGT], or total bilirubin), immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal condition, or other major disease.
4. The subject had a history of any malignant disease.
5. The subject had a history of more than one herpes zoster episode or multidermatomal herpes zoster.
6. The subject had a history of an opportunistic infection (e.g. cytomegalovirus, pneumocystis carinii, aspergillosis, clostridium difficile).
7. The subject had a history of or ongoing chronic or recurrent infectious disease (e.g. infected indwelling prosthesis, osteomyelitis, chronic sinusitis).
8. The subject had major trauma or surgery in the 2 months before screening or at any time between screening and check-in.
9. The subject had an acute infection within 2 weeks before screening or at any time between screening and check-in including, but not limited to, history, signs, or symptoms of a common cold (eg, mild rhinorrhea), untreated oral/dental abnormalities (e.g. untreated dental caries as determined by examination of the mouth), or untreated disruption of the skin.
10. The subject had clinically significant abnormal ECG findings at screening, check-in visits, or predose, as determined by the Investigator.
11. The subject had a supine blood pressure measurement outside the ranges of 90 to 140 mm Hg systolic or 45 to 90 mm Hg diastolic (measured after a rest of at least 5 minutes) at screening, check-in, or predose. Note: If either value was out of the range, blood pressure measurements may be repeated in the supine position at intervals of 5 to 10 minutes up to 3 times. If the mean systolic or diastolic measurement continues to exceed the stated limits, the subject will be excluded.
12. The subject had a pulse of fewer than 45 beats per minute (bpm) or greater than 100 bpm(measured after a rest of at least 5 minutes) at screening, check-in, or predose.
13. The subject tests positive for tuberculosis (TB) at screening by the QuantiFERON-TB Gold Test, or has a history of latent, inadequately treated, or active TB.
14. The subject had a known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) types 1 or 2 at screening.
15. The subject had used prescription or over-the-counter (OTC) medication (other than ≤2 g/day paracetamol [acetaminophen] or ≤800 mg/day ibuprofen), vitamins, or herbal remedies, within 2 weeks or 5 half-lives before study drug administration, whichever was longer.
16. The subject had participated in another clinical study of a new investigational drug or has received an investigational drug within the 3 months or 5 half-lives (if available) before study drug administration, whichever is longer.
17. The subject had a loss of more than 400 mL of blood (e.g. a blood donation) within 2 months before study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before check-in, or plans to donate blood during the study or within 3 months after the study.
18. The subject had a history of alcohol abuse (defined as an alcohol intake more than 21 units per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 240 mL of beer, 120 mL of wine, or 1 single shot of spirits. The subject will be required to abstain from alcohol consumption 48 hours prior to screening or check-in.
19. The subject was a current smoker or has a history of smoking.
20. The subject had a positive test for alcohol or drugs of abuse (barbiturates, methamphetamine, benzodiazepines, morphine/opiates, phencyclidine (PCP), amphetamines, tetrahydrocannabinol (THC), methylenedioxymethamphetamine (MDMA), cocaine, methadone, and cotinine) at screening or check-in.
21. The subject was unable to participate in, or successfully complete, the study, in the opinion of their general practitioner or the investigator, because the subject was any of the following:

    1. mentally or legally incapacitated, or unable to give consent for any reason
    2. in custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitarium or social institution
    3. unable to be contacted in case of emergency
    4. unlikely to cooperate or comply with the clinical study protocol or was unsuitable for any other reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
After single ascending doses, number of subjects with treatment-emergent adverse events (TEAEs) after dosing with EI-1071 | Up to 7 days
  Experience at least 1 treatment-emergent adverse event
After multiple ascending doses, number of subjects with TEAEs after dosing with EI-1071 | Up to 21 days
  Experienced at least 1 treatment-emergent adverse event
After multiple ascending doses, number of subjects with adverse events (AEs) leading to discontinuation in the EI-1071 cohorts. | Up to 14 days
  Discontinued due to adverse event

SECONDARY OUTCOMES:
Cmax | Single dose: up to 48 hours; Multiple dose: up to 16 days
  Maximum observed serum concentration
Tmax | Single dose: up to 48 hours; Multiple dose: up to 16 days
  Time to reach Cmax
t1/2 | Single dose: up to 48 hours; Multiple dose: up to 16 days
  Terminal half-life
AUC-last | Single dose: up to 48 hours; Multiple dose: up to 16 days
  Area under the curve from the time of dosing to the time of the last measurable concentration
AUC-inf | Single dose: up to 48 hours; Multiple dose: up to 16 days
  Area under the curve from the time of dosing extrapolated to infinity
Colony Stimulating Factor 1 (CSF1) concentration in blood after multiple-dose administration | Up to 15 days
  Amount of Colony Stimulating Factor 1
Monocyte count in blood after multiple-dose administration | Up to 15 days
  Count of monocyte subsets

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yun Pai, Study Director — Elixiron Inc.
Locations (1):
- Parexel Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No